CLINICAL TRIAL: NCT01612624
Title: FACIAL AND HAND ANALYSIS, SLEEP APNEA AND SPEECH IN PATIENTS WITH ACROMEGALY: A PROSPECTIVE STUDY TO INVESTIGATE CHANGES IN CRANIOFACIAL AND HAND CHARACTERISTICS, SLEEP APNEA AND SPEECH DURING TREATMENT AND AFTER REMISSION
Brief Title: Prospective Study on Changes in Acromegaly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: AP1
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Rationale: Acromegaly is the clinical syndrome that results from an excess of growth hormone (GH). Craniofacial and hand disproportions due to soft tissue swelling and new bone formation are highly prevalent in patients with active acromegaly. Besides the cosmetic aspects, these changes can impair the quality of life because of the significant morbidity with respect to oral, maxillofacial and hand pathologies as well as respiratory problems such as sleep apnea and changes in speech. At present it is unclear if these craniofacial and hand disproportions, sleep apnea and speech changes are (partially) reversible after successful treatment. Therefore there is no consensus about the information patients should be given about (partial) recovery of facial and hand disproportions after treatment and how the follow-up with respect to oral, maxillofacial, respiratory and hand pathology should be organized. Facial and hand analysis using a 3D stereophotograph and a 3D fusion model of a 3D stereophotograph and a 3D skull reconstruction via cone beam computed tomography (CT)-scan makes it possible to investigate the craniofacial changes due to acromegaly in all facial dimensions together (dentition, bone and soft tissue) and the relational proportions between these facial structures. 3D stereophotography can do the same for the soft tissues of the hand. Combined with disease specific and general quality of life (QOL) questionnaires, a correlation between quality of life and craniofacial and hand disproportions can be determined. Combined with sleep- and speech analysis, a correlation between sleep apnea, speech and craniofacial disproportions can be determined.

Primary objective: To investigate the changes in facial- and hand analysis in patients with acromegaly as a result of medical treatment and pituitary surgery, and to investigate the changes in relational proportions between facial- and hand structures, incidence and severity of sleep apnea, incidence and severity of speech changes and QOL.

Study design: a prospective case-control study. Study population: Approximately thirty patients newly diagnosed with acromegaly . The results of facial and hand analysis, sleep apnea research and speech analysis of the patient group in different phases of the disease will be compared to the results of a healthy control group.

Main study parameters/endpoints: Parameters of facial analysis with 3D stereophotography and cone beam CT and hand analysis with 3D stereophotography , biochemical parameters of disease activity, disease related QOL assessed by 2 validated QOL questionnaires (,the AcroQol and RAND-36 ), speech analysis, the results of the voice handicap index questionnaire and severity of sleep apnea assessed by complete overnight polysomnography and the Epworth sleepiness scale questionnaire.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: As a result of participating in this study, subjects have to undergo a cone beam CT. The cone beam CT is associated with exposure to X-ray radiation of 0.069-0.135mSv. This is the same amount of radiation as the amount of background radiation that each person receives in 7 days time during daily life. No adverse effects are expected from this amount of exposure. The investigations will take 10-70 minutes adjacent to every regular outpatient clinic visit. In addition , for polysomnography, subjects will be investigated overnight one or three times in 2,5 years, depending on the results of the first screening polysomnography.

Assessment of changes in body appearance, sleep disturbances, speech changes and QOL in a prospective longitudinal fashion will increase the knowledge of the impact of the disease on patient perception of well-being and functioning and will help us refine the treatment goals in patients with acromegaly

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed acromegaly
* Diagnosis is biochemically confirmed by an increased IGF-1 level (> mean +2 standard deviations for age) and insufficient suppression of serum GH levels (e.g. GH levels ≥ 2mU/l) during oral glucose tolerance test.
* Subjects should be over 18 years old with the ability to read and comprehend the Dutch language

Exclusion Criteria:

4.3 Exclusion criteria imaging face:

* Pregnancy
* Maxillofacial surgical treatment in the past.

Exclusion criteria 3D imaging of the hand:

* Hand surgery in the past

Exclusion criteria Speech analysis:

* Speech pathology unrelated to acromegaly

Exclusion criteria polysomnography:

* Co-morbidities that could influence the prevalence of sleep apnea (e.g. muscular dystrophy, known hypothyroidism)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acromegaly patients and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-05

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Gelderland, Netherlands